CLINICAL TRIAL: NCT03836001
Title: A Neurokinin-1 Receptor Antagonist for the Treatment of Pruritus in Patients With Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Epidermolysis Bullosa Research Partnership (Other Government); Vyne Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Albert Chiou, Assistant Professor of Dermatology., Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49084
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — serlopitant; Sugars

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, single-center, randomized, double-blind, placebo-controlled, parallel-arm trial evaluating the effects of serlopitant at 5 mg by mouth daily on EB-related itch.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Participants will undergo two months of dosing with a placebo (inactive drug or sugar pill), followed by one month of washout. After the washout period, all participants were invited to participate in an open-label extension study with serlopitant 5 mg daily. The duration of the open-label extension study was either 12 months (for those who enrolled before May 2020) or 3 months (for those who registered after May 2020) due to drug availability.
  Interventions: Drug: Placebo Oral Tablet
- Serlopitant Tablet (Active Comparator): Participants will undergo two months of Serlopitant 5mg daily per oral, followed by one month of washout. After the washout period, all participants were invited to participate in an open-label extension study with serlopitant 5 mg daily. The duration of the open-label extension study was either 12 months (for those who enrolled before May 2020) or 3 months (for those who registered after May 2020) due to drug availability.
  Interventions: Drug: Serlopitant Tablet

INTERVENTIONS:
Drug: Serlopitant Tablet — Serlopitant is a small molecule, highly selective NK1-R (neurokinin-1 receptor) antagonist. Two critical mediators of the urge to scratch are Substance P, or SP, and its receptor, NK1-R. SP is a naturally occurring peptide in the tachykinin neuropeptide family. Tachykinins have a broad range of functions in the nervous and immune systems. SP binding of NK1-R has been shown to be a key mediator of sensory nerve signaling, including the itch-scratch reflex and the vomiting reflex.
  Other Names: VPD-737
  Arms: Serlopitant Tablet
Drug: Placebo Oral Tablet — The placebo is a tablet that looks like a drug but has no drug or other active ingredient in it.
  Other Names: Sugar pill
  Arms: Placebo Oral Tablet

SUMMARY:
To determine if Serlopitant (when taken by mouth) is safe and works on itch in patients aged 13 and above with EB.

DETAILED DESCRIPTION:
The investigator will determine whether more patients taking serlopitant 5 mg daily as compared to placebo can achieve at least a 3-point reduction in the 24-hour Average Itch Numeric Rating Scale (NRS) following two months of treatment.

Secondary objectives include;

1. comparative weekly change in daily worst itch NRS,
2. comparative weekly change in daily average itch NRS,
3. the proportion of patients who achieve at least 30% or 50% reduction in Average Itch NRS at month 2,
4. proportion of patients achieving 2-point and 4-point reductions in Average Itch NRS at month 2,
5. Patient Global Impression of Change (PGIC) at month 2, the change in participant static assessment of itch at month 2, and
6. assessment of the safety of serlopitant in adolescents (≥13 y.o.) and adults with epidermolysis bullosa-related itch.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are at least 13 years of age.
2. Willing and able to understand and sign informed assent/consent. Adolescents will need a parent or guardian willing and able to give consent.
3. Clinical diagnosis of epidermolysis bullosa (dystrophic, junctional or simplex).
4. History of chronic pruritus of at least 6 weeks in duration
5. On the Screening Visit or Screening phone call, patients must have an NRS pruritus score of at least 5 on average itch score in the past 24 hours
6. Female subjects must be of non-childbearing potential (ie, post-menopausal for at least 1 year, had a hysterectomy, or had a tubal ligation) or, if of childbearing potential, must have a confirmed negative urine pregnancy test prior to study treatment and be willing to use effective contraception for the duration of the trial. Effective contraception is defined as follows: oral/implant/injectable/ transdermal contraceptives, intrauterine device, condom with spermicide, or diaphragm with spermicide. Abstinence or partner's vasectomy is acceptable if the female agrees to use effective contraception if she decides to discontinue abstinence or to have sexual intercourse with a non-vasectomized partner.
7. Judged to be in good health based upon the results of a physical examination, medical history, and safety laboratory tests.

Exclusion Criteria:

1. Have any medical condition or disability that would interfere with the assessment of safety or efficacy in this trial or would compromise the ability of the subject to travel to Stanford or to undergo study procedures or to give informed consent.
2. Have a history of sensitivity to any components of the study material.
3. Are females of childbearing potential who are unwilling to use adequate contraception or who are breast feeding.
4. Have any chronic or acute medical condition that, in the opinion of the investigator, might interfere with the study results or place the subject at undue risk.
5. Have chronic renal disease, i.e., serum creatinine greater than 2 times the upper limit of normal.
6. Have chronic liver disease. Subjects with hepatitis B and C who have normal liver function may be enrolled.
7. Have a current malignancy (such as Hodgkin's lymphoma, B or T cell lymphoma, or myeloma) or blood cell dyscrasia (e.g., polycythemia or myelofibrosis) that would lead to systemic chronic pruritus.
8. Have a history of thyroid cancer, thyroid nodules, inadequately treated thyroid disease, or abnormal TSH or free T4 at screening.
9. Have a history of abnormalities in adrenal or pituitary function (pituitary adenoma, adrenal insufficiency, or adrenal nodule).
10. Screening cortisol level < 3 mcg/dL
11. Unevaluated abnormalities in cortisol, ACTH, or prolactin.
12. Have pruritus of psychogenic etiology (delusions of parasitosis, obsessive compulsive disorder and major depression) or neuropathic etiology (due to shingles, spinal cord injury or with neurologic deficit).
13. Have pruritus due to urticaria, drug allergy, or infection (such as pityriasis rosacea or tinea or active human immunodeficiency virus [HIV]). Note: Subjects with HIV who have undetectable viral load, and stable retro-viral therapy may enroll.
14. Have taken investigational medications within 30 days prior to Screening.
15. Are unwilling to discontinue specific medications that, in the view of the investigator may have significant interactions with the trial drug, for at least two weeks prior to initiation of study and throughout the study period (this includes miconazole, delavirdine, conivaptan, Clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir).
16. Are unable or unwilling to maintain their current anti-itch and opioid-based pain medications at a stable dosage through the course of the two months of active treatment (including but not limited to opioid pain medications, antihistamines, and gabapentin)
17. Started or changed medications, creams, or emollients including over-the-counter (OTC) preparations or bath oil treatment specifically for relief of pruritus within 30 days prior to Screening.
18. Within in the past 12 months, have expressed suicidal ideation with some intent to act.
19. Have any social or medical condition (e.g. alcoholism, drug dependency, psychotic state) that, in the investigator's opinion, might interfere with the subject's ability to comply with the requirements of the protocol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Chiou, MD/MBA, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiou AS, Choi S, Barriga M, Dutt-Singkh Y, Solis DC, Nazaroff J, Bailey-Healy I, Li S, Shu K, Joing M, Kwon P, Tang JY. Phase 2 trial of a neurokinin-1 receptor antagonist for the treatment of chronic itch in patients with epidermolysis bullosa: A randomized clinical trial. J Am Acad Dermatol. 2020 Jun;82(6):1415-1421. doi: 10.1016/j.jaad.2019.09.014. Epub 2019 Sep 18. PMID 31541747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants were consented but failed initial screening and were not allocated to treatment. Two participants failed initial screening but were re-screened and entered the study.
  A protocol amendment in May 2020 changed the duration of the follow-up period from 12 months to 3 months.
Groups:
- Placebo Oral Tablet: Patients undergo two months of dosing with placebo followed by one month of wash-out. All patients may continue in a 3-month open label extension with serlopitant at 5 mg (taken by mouth) daily for continued safety monitoring.
- Serlopitant Tablet: Patients who will undergo two months of Serlopitant dosing, followed by one month of wash-out. All patients may continue in a 3-month open label extension with serlopitant at 5 mg (taken by mouth) daily for continued safety monitoring.
- Open-label Extension: 3-month open label extension with serlopitant at 5 mg (taken by mouth) daily for continued safety monitoring.
Period: Blinded Phase (2 Months)
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet | Open-label Extension
Started | 12 | 12 | 0
Completed | 12 | 10 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Washout (1 Month)
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet | Open-label Extension
Started | 12 | 10 | 0
Completed | 12 (6 participants continued into the open label extension.) | 10 (4 participants continued into the open label extension.) | 0
Not Completed | 0 | 0 | 0
Period: Open-label Extension (3 or 12 Months)
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet | Open-label Extension
Started | 0 | 0 | 10
Entered 12-month Follow-up Period | 0 | 0 | 2
Entered 3-month Follow-up Period | 0 | 0 | 8
Completed | 0 | 0 | 8
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Enrolled in other clinical study | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 67] | 22 [13 to 73] | 31 [13 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 6 | 14
  Asian | 3 | 0 | 3
  African American | 0 | 1 | 1
  Other | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24
Epidermolysis Bullosa (EB) Subtype [Count of Participants; unit: Participants]
  EB simplex | 2 | 1 | 3
  Junctional EB | 1 | 0 | 1
  Dominant dystrophic EB | 1 | 2 | 3
  Recessive dystrophic EB | 8 | 9 | 17
Average Itch Numeric Rating Scale (AI-NRS) [Median (Full Range); unit: score on a scale] — Scale range: 0 to 10, higher scores mean more itch.
  score on a scale | 6 [2 to 8] | 7 [1 to 9] | 6 [1 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve at Least a 3-point Reduction in AI-NRS.
Description: Participants will be asked to complete a daily itch diary with their average itch numeric rating scale (AI-NRS) over the past 24 hours. Score range: 0 to 10, higher scores mean more itching.
Time Frame: baseline and after two months of treatment
Population: Data were analyzed using the last observation carried forward method (LCOF)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
Participants | 1 | 3
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; Test type: Superiority; p = 0.59, Fisher Exact — A p-value of <0.05 would be considered statistically significant

2. Secondary Outcome: Number of Patients Who Achieve at Least a 2-point Reduction in AI-NRS.
Description: as for outcome 1
Time Frame: baseline and after two months of treatment
Population: Data were analyzed using the last observation carried forward method (LCOF)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
Participants | 2 | 3
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; Test type: Superiority; p = 1, Fisher Exact — A p-value of <0.05 would be considered statistically significant

3. Secondary Outcome: Number of Patients Who Achieve at Least a 4-point Reduction in AI-NRS.
Description: as for outcome 1
Time Frame: baseline and after two months of treatment
Population: Data were analyzed using the last observation carried forward method (LCOF)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
Participants | 1 | 1
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; Test type: Superiority; p = 1, Fisher Exact — A p-value of <0.05 would be considered statistically significant

4. Secondary Outcome: Number of Patients Who Achieve at Least a 30% Reduction in AI-NRS.
Description: as for outcome 1
Time Frame: baseline and after two months of treatment
Population: Data were analyzed using the last observation carried forward method (LCOF)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
Participants | 4 | 3
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; Test type: Superiority; p = 0.67, Fisher Exact — A p-value of <0.05 would be considered statistically significant

5. Secondary Outcome: Number of Patients Who Achieve at Least a 50% Reduction in AI-NRS.
Description: as for outcome 1
Time Frame: baseline and after two months of treatment
Population: Data were analyzed using the last observation carried forward method (LCOF)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
Participants | 1 | 1
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; Test type: Superiority; p = 1, Fisher Exact — A p-value of <0.05 would be considered statistically significant

6. Secondary Outcome: Weekly Worst Itch NRS
Description: Participants will be asked to complete a daily itch diary with their worst itch numeric rating scale (WI-NRS) over the past 24 hours. Score range: 0 to 10, higher scores mean more itching.
Time Frame: baseline and week 1, 2, 3, 4, 5, 6, 7, and 8
Population: Daily diary data were averaged weekly. The missing weekly data have been imputed by the mean WI-NRS value of each participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
score on a scale
  baseline | 6.1 (2.3) | 7.3 (1.6)
  week 1 | 6.0 (2.3) | 6.3 (1.7)
  week 2 | 6.1 (2.0) | 5.9 (1.6)
  week 3 | 6.5 (1.9) | 5.7 (1.8)
  week 4 | 6.4 (1.7) | 5.6 (2.0)
  week 5 | 6.4 (2.2) | 5.7 (2.2)
  week 6 | 6.0 (2.3) | 5.8 (2.1)
  week 7 | 6.0 (2.2) | 5.6 (2.2)
  week 8 | 6.0 (2.4) | 5.4 (2.1)
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; Analysis of change from baseline through week 8 including all time points. For this analysis, data were censored at the time of participant discontinuation; Test type: Other; p = 0.09, Mixed Models Analysis — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.24 to 0.02]

7. Secondary Outcome: Weekly AI-NRS
Description: as for outcome 1
Time Frame: baseline and week 1, 2, 3, 4, 5, 6, 7, and 8
Population: Daily diary data were averaged weekly. The missing weekly data have been imputed by the mean AI-NRS value of each participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
score on a scale
  baseline | 5.3 (2.2) | 6.3 (2.3)
  week 1 | 5.1 (2.2) | 5.6 (2.2)
  week 2 | 5.3 (1.9) | 5.6 (1.9)
  week 3 | 5.5 (2.0) | 5.2 (2.4)
  week 4 | 5.4 (1.7) | 5.2 (2.2)
  week 5 | 5.2 (2.0) | 5.1 (2.4)
  week 6 | 5.0 (2.1) | 5.1 (2.6)
  week 7 | 4.8 (1.7) | 5.2 (2.7)
  week 8 | 4.8 (2.0) | 5.0 (2.7)
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.16, Mixed Models Analysis — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.19 to 0.03]

8. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: PGIC categorized as "Very much better", "Moderately better", "A little better", "No change", "A little worse", "Moderately worse", and "Very much worse".
Time Frame: month 2
Population: Participants who completed the month 2 assessment are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 10
Participants
  Very much better | 0 | 2
  Moderately better | 1 | 0
  A little better | 5 | 3
  No change | 5 | 5
  A little worse | 0 | 0
  Moderately worse | 1 | 0
  Very much worse | 0 | 0

9. Post Hoc Outcome: Dressing/Bathing NRS
Description: Participants will be asked to complete a daily itch diary with their itch Numeric Rating Scale (NRS) during dressing/bathing. Score range: 0 to 10, higher scores mean more itching.
Time Frame: baseline and week 1, 2, 3, 4, 5, 6, 7, and 8
Population: Daily diary data were averaged weekly. The missing weekly data have been imputed by the mean Dressing/Bathing-NRS value of each participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 12 | 12
score on a scale
  baseline | 5.3 (2.6) | 6.8 (3.1)
  week 1 | 5.1 (2.3) | 5.7 (3.0)
  week 2 | 5.0 (2.1) | 6.0 (2.8)
  week 3 | 5.5 (2.5) | 5.4 (3.1)
  week 4 | 5.4 (2.7) | 5.1 (3.1)
  week 5 | 5.6 (2.6) | 5.5 (2.9)
  week 6 | 5.6 (2.7) | 5.5 (3.2)
  week 7 | 5.6 (2.8) | 5.4 (3.2)
  week 8 | 5.3 (2.7) | 5.4 (3.2)
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Serlopitant Tablet; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.002, Mixed Models Analysis — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.41 to -0.09]

10. Secondary Outcome: Change in Static Participant Assessment of Itch
Description: Severity of itch over past 7 days assessed as Very Severe, Severe, Moderate, Mild, or None.
  Change is reported as the number of participants with 3-category improvement, 2-category improvement, 1-category improvement, no change, or worse.
Time Frame: month 2
Population: Participants who enrolled after protocol amendment adding this outcome measure are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet
Number analyzed (Participants) | 5 | 4
Participants
  3-category improvement | 0 | 1
  2-category improvement | 0 | 1
  1-category improvement | 2 | 0
  No change | 3 | 2
  Worse | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 15 months
Groups:
- Placebo Oral Tablet: Patients undergo two months of dosing with a placebo followed by one month of wash-out. All patients were invited to participate in an open-label extension study.
- Serlopitant Tablet: Patients who will undergo two months of Serlopitant dosing, followed by one month of wash-out. All patients were invited to participate in an open-label extension study.
- Open-label Extension: Participants took oral serlopitant 5mg daily for either 12 months (for those who enrolled before May 2020) or 3 months (for those who registered after May 2020).
Arm/Group | Placebo Oral Tablet | Serlopitant Tablet | Open-label Extension
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/12 | 0/10
Other Adverse Events (participants affected / at risk) | 9/12 | 10/12 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Oral Tablet (N=12) | Serlopitant Tablet (N=12) | Open-label Extension (N=10)
Wound infection (Infections and infestations) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Bacteremia (sepsis) (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Oral Tablet (N=12) | Serlopitant Tablet (N=12) | Open-label Extension (N=10)
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Soft stool (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Elevated ALT (Hepatobiliary disorders) | 0 | 1 | 0
Elevated GGT (Hepatobiliary disorders) | 0 | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Elevated prolactin (Investigations) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Fatigue (General disorders) | 1 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic headaches (Nervous system disorders) | 0 | 1 | 0
Type 2 diabetes (Endocrine disorders) | 0 | 1 | 0
Corneal abrasion (Eye disorders) | 0 | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swollen cheek due to wound (Infections and infestations) | 0 | 1 | 0
Flu-like symptoms (General disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Enlarged lymph nodes (Blood and lymphatic system disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0
Worsening anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Cracked tooth (Gastrointestinal disorders) | 0 | 1 | 0
Inflamed cyst (General disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Irritant dermatitis around G-tube (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hematuria (Blood and lymphatic system disorders) | 0 | 2 | 0
Kidney stone surgery (Renal and urinary disorders) | 0 | 1 | 0
Microscopic pyuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
The COVID-19 infection (Infections and infestations) | 0 | 0 | 2
Enlarged parotid gland (Blood and lymphatic system disorders) | 0 | 1 | 0
Elevated leukocyte esterase (Blood and lymphatic system disorders) | 1 | 0 | 0
Pruritus of pharynx (Gastrointestinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The primary limitation of the study is the small sample size due to the rarity of EB, the COVID-19 pandemic-related disruptions, and limited drug availability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT03836001/Prot_SAP_000.pdf